CLINICAL TRIAL: NCT07026565
Title: Psychotherapy Group for Parents of Children With Leber Congenital Amaurosis
Brief Title: Psychotherapy Group for Parents of Children With LCA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Genética Ocular (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: InstitutoGeneticO
Record Dates: First submitted 2025-03-28; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Leber Congenital Amaurosis (LCA)
Keywords: psychotherapeutic group; Leber congenital amaurosis; Acceptance and Commitment Therapy; Parental psychological well-being
MeSH Terms: conditions — Leber Congenital Amaurosis | interventions — Psychotherapy, Group; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The psychotherapy group will consist of 10 virtual sessions, each lasting 1 hour and 15 minutes. Each session will begin with a mindfulness exercise to bring the participants into the present moment, followed by a pre-determined topic for discussion. At the end of each session, there will be a closing segment to summarize the reflections and teachings of the day, and a homework assignment will be provided. The topics covered will be: Opening, Psychoeducation, Diagnosis Report, Acceptance, Psychological Flexibility, Cognitive Defusion, Self as Context, Values, Committed Action, and Closure.
  Interventions: Behavioral: Psychotherapy group for parents
- Control Group (Active Comparator): For the parents who will participate in the control group, the steps undertaken will include the administration of the Self-Reporting Questionnaire, Parental Stress Scale, Acceptance and Action Questionnaire, Cognitive Fusion Questionnaire, and Freiburg Mindfulness Inventory, before the intervention, after the intervention, and after 3 months.
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: Psychotherapy group for parents — The psychotherapy group will consist of 10 virtual sessions, each lasting 1 hour and 15 minutes. Each session will begin with a mindfulness exercise to bring the participants into the present moment, followed by a pre-determined topic for discussion. At the end of each session, there will be a closing segment to summarize the reflections and teachings of the day, and a homework assignment will be provided. The topics covered will be: Opening, Psychoeducation, Diagnosis Report, Acceptance, Psychological Flexibility, Cognitive Defusion, Self as Context, Values, Committed Action, and Closure.
  Arms: Intervention Group
Behavioral: Control Group — For the parents who will participate in the control group, the steps undertaken will include the administration of the Self-Reporting Questionnaire, Parental Stress Scale, Acceptance and Action Questionnaire, Cognitive Fusion Questionnaire, and Freiburg Mindfulness Inventory, before the intervention, after the intervention, and after 3 months.
  Arms: Control Group

SUMMARY:
The objectives of this study are to evaluate the effect of a group psychotherapy intervention for parents of children/adolescents with LCA on indicators of emotional health, parental stress, acceptance, cognitive defusion, and mindfulness. The study design is a repeated measures design with pre-, post-, and 3-month follow-up assessments. Forty parents of children and adolescents with LCA will be included in the sample. Twenty will participate in the psychotherapy groups, divided into 2 groups of 10 people, and 20 will be in the control group. To assess the indicators mentioned in the objective, the following questionnaires will be applied: Self-Reporting Questionnaire, Parental Stress Scale, Acceptance and Action Questionnaire, Cognitive Fusion Questionnaire, and Freiburg Mindfulness Inventory. A subsequent data analysis will be conducted to evaluate and correlate these indicators before, after, and 3 months post-intervention.

DETAILED DESCRIPTION:
INTRODUCTION

Parent-Child Relationships and Their Influence on Child Development:

Families with children diagnosed with inherited retinal diseases (IRD) exhibit high levels of depression, anxiety, and social isolation. Additionally, parents of children with IRD experience financial stress, as their productivity is affected by caregiving responsibilities, alongside increased expenditures on general health and rehabilitation. Regarding Leber congenital amaurosis (LCA), there are no studies assessing these indicators. However, since LCA falls under the IRD category, it can be presumed to have similar effects.

The parent-child relationship in the context of autism spectrum disorder (ASD) is frequently associated with high levels of parental stress and psychological distress. Previous studies have identified maladaptive behavior in children with ASD, particularly problematic behaviors, as the primary factor increasing parental stress, negatively affecting their mental health and psychological adjustment. Coping strategies, such as experiential avoidance, often linked to mental health issues, exemplify how parents may be negatively impacted by the complexity of their children's behavior.

Other studies investigating the emotional health of parents of children with various chronic illnesses have reported similar findings, indicating that experiential avoidance is directly related to parental psychological distress. Experiential avoidance refers to passivity towards a behavior or even fleeing from it. The mechanism that should replace experiential avoidance is psychological acceptance. Acceptance is a process that involves consciously embracing difficult situations without attempting to suppress or avoid them. It benefits individuals who need to accept immutable conditions, such as chronic, incurable, or untreatable health conditions.

Psychological acceptance has been studied among parents of children with intellectual disabilities. A study analyzed the adaptation of mothers of children with intellectual disabilities and observed that psychological acceptance was inversely related to maternal anxiety, stress, and depression. A more recent study, found that psychological acceptance partially mediated the relationship between the child's problematic behavior and parental stress, depression, and anxiety. Problematic behaviors were linked to reduced psychological acceptance, which, in turn, was associated with increased parental maladjustment.

Acceptance and Commitment Therapy (ACT) incorporates the concepts of experiential avoidance and acceptance as core elements. As a third-wave behavioral therapy, ACT is grounded in functional contextualism and informed by Relational Frame Theory (RFT). Unlike therapeutic models that prioritize symptom reduction, ACT considers this reduction as a side effect, focusing primarily on the development of psychological flexibility (PF).

PF is a transdiagnostic concept, typically represented by the "Hexaflex" diagram, which outlines six fundamental, interconnected processes considered essential for psychological well-being:

Acceptance: Recognizing and embracing internal experiences (such as emotions, feelings, thoughts, and memories) without attempting to avoid or modify them, cultivating a curious and interested attitude.

Cognitive Defusion: The ability to distance oneself from thoughts and feelings, perceiving them as subjective internal events rather than absolute realities, fostering an observational stance regarding cognitions and their effects on behavior.

Flexible Attention: Cultivating awareness of the impermanence of internal and external occurrences, recognizing moment-to-moment changes.

Self-as-Context: Encouraging individuals to recognize stable and transient aspects of the "self." While emotions and thoughts shift according to context, the perspective (or self) from which these events are observed remains constant.

Committed Action: Identifying and carrying out actions aligned with one's values and life goals, even when facing emotional and cognitive discomfort.

Values: Exploring and identifying fundamental principles, such as honesty and courage, that transcend specific goals and guide a meaningful and coherent life.

Given the high level of psychological distress experienced by parents of children with ASD, intellectual disabilities, or chronic illnesses, various psychotherapy initiatives have been developed to improve this condition. A review examined evidence on psychological interventions to reduce stress in parents of children with intellectual disabilities, emphasizing group cognitive-behavioral techniques, which have proven particularly effective in alleviating parental distress, with a greater effect on mothers. One study developed a group psychotherapy program based on ACT to reduce distress in parents of children with life-threatening illnesses. Its results showed significant reductions in post-traumatic stress symptoms, as well as improvements in psychological flexibility and mindfulness. Lastly, a study conducted a two-day ACT training workshop for parents of children with ASD. This training, based on the six pillars of ACT, led to improvements in parental emotional health and a reduction in experiential avoidance.

To date, no studies have evaluated psychotherapeutic interventions for parents of children with LCA. However, it is assumed that these parents experience psychological distress, as LCA is also a chronic disease, and IRD, as previously mentioned, causes emotional suffering in parents. Therefore, group psychotherapy initiatives based on ACT could help improve these individuals' emotional health.

OBJECTIVE

To evaluate the effect of a group psychotherapy intervention for parents of children/adolescents with LCA on indicators of emotional health, parental stress, acceptance, cognitive defusion, and mindfulness.

1. To assess emotional health, parental stress, acceptance, cognitive defusion, and mindfulness in parents of children/adolescents with LCA before the intervention.
2. To evaluate the impact of the intervention on emotional health, parental stress, acceptance, cognitive defusion, and mindfulness in parents of children/adolescents with LCA immediately after and three months post-intervention.

METHOD

This study will evaluate the efficacy of a psychotherapy group in enhancing emotional health, acceptance, mindfulness, cognitive defusion, and reducing parental stress. A repeated-measures design with pre-, post-, and three-month follow-up assessments was utilized. The intervention consists of 10 virtual sessions lasting 1 hour and 15 minutes, guided by ACT-compatible principles. This study was approved by the UNIFESP Research Ethics Committee (approval number 6.260.956). The psychologists responsible for the group, CFCV and LFF, are ACT specialists, with the former being diagnosed with LCA.

Sample

Forty parents of children and adolescents with LCA will be included. Twenty will participate in psychotherapy groups, and twenty will be in the control group. Parents with diagnosed mental disorders prior to their child's birth and unrelated to LCA acceptance will be evaluated by psychologists and excluded from the sample. Exclusion criteria were established based on the impact of these variables on the study's analysis. Initially, parents undergoing individual psychotherapy and/or psychiatric medication use will be excluded.

Intervention: Psychotherapy Group

The psychotherapy group will consist of 10 virtual sessions of 1 hour and 15 minutes. Each session will begin with a mindfulness exercise to anchor participants in the present moment, followed by a discussion of a pre-determined theme. At the end of each session, a closing discussion will summarize key insights and assign a take-home activity. Table 1 outlines the psychotherapy group plan.

This Psychotherapy Group model was created by the author CFCV, and this ACT-based intervention was referenced from Hayes et al.

Procedures

Parents will be invited to participate in the psychotherapy group through phone contact from the Instituto de Genética Ocular in January 2025. Subsequently, psychologists CFCV and LFF will conduct 30-minute screenings for each participant. Five assessments (SRQ-20, EEPa, AAQ-II, CFQ, and FMI) will be administered in the following session, lasting 1 hour. Weekly sessions will take place from February to April 2025 via Google Meet. Assessments will be re-administered in May 2025, with a final follow-up in August 2025.

Data Analysis The collected data will be analyzed using the R statistical software, version 4.4.1. Descriptive analyses will be performed, including calculations of mean, mode, median, standard deviation, and percentiles. Inferential analysis will also be conducted using Fisher's exact test, Wilcoxon test, Student's t-test (independent and paired), as well as normality (Shapiro-Wilk), homogeneity (Levene), and sphericity (Mauchly) tests. The statistical significance level was set at 5% (p=0.05).

ELIGIBILITY:
Inclusion Criteria:

* Forty parents of children and adolescents with LCA will be included in the sample. These parents must have both the clinical and genetic diagnoses of their children.

Exclusion Criteria:

* Parents with diagnosed mental disorders prior to the birth of their children and unrelated to the acceptance of LCA will be evaluated by the psychologists and excluded from the sample. The exclusion criteria were assigned based on the impact of these variables on the study analysis. Additionally, parents who are undergoing individual psychotherapy and/or using psychiatric medication will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-02-27 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Self-Reporting Questionnaire | 2 Months
  The SRQ-20 questionnaire has been validated for the Brazilian population and contains 20 items that assess the presence or absence of mental disorders. The questions are scored in a dichotomous format, and a score of 7 or more indicates the possible presence of a mental disorder. The SRQ-20 serves as a screening tool but does not identify the specific mental disorder experienced by the patient.
Freiburg Mindfulness Inventory | 2 Months
  The FMI assesses mindfulness through 14 items and has been validated for the Brazilian population. Each item is rated on a Likert scale from 1 to 4. Higher scores indicate that the individual acts more consistently with mindfulness.
Cognitive Fusion Questionnaire | 2 Months
  The CFQ is a tool used to assess the degree of cognitive fusion, which refers to the tendency of individuals to identify with their thoughts and treat them as absolute truths. It consists of 7 items, is validated for use with the Brazilian population, and responses are rated on a scale from 1 to 7. Higher scores indicate a higher level of cognitive fusion.
Acceptance and Action Questionnaire | 2 Months
  The AAQ-II questionnaire has been validated and adapted for Portuguese and contains 7 items that assess inflexible behaviors. The items are rated on a Likert scale from 1 to 7, where 1 means "Never" and 7 means "Always." Lower scores indicate greater psychological flexibility, meaning a higher ability to deal with different events in different ways.
Parental Stress Scale | 2 Months
  The EEPa has been validated and adapted for Brazil and contains 16 items-eight questions related to parental satisfaction with the parenting experience and eight related to parental stressors. Responses are given on a Likert scale from 0 (strongly disagree) to 4 (strongly agree). The total score is 64 points, and higher scores indicate greater levels of parental stress experienced by participants.

CONTACTS AND LOCATIONS:
Overall Officials: Cecília F Vasconcellos, PhD studant, Principal Investigator — Ocular Genetic Institute; JULIANA F SALLUM, Post-doc, Study Chair — Ocular Genetic Institute; Caio Marques, PhD studant, Study Director — Ocular Genetic Institute
Locations (1):
- Instituto de Genética Ocular, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-17): https://cdn.clinicaltrials.gov/large-docs/65/NCT07026565/Prot_SAP_000.pdf
  • Informed Consent Form (2024-07-17): https://cdn.clinicaltrials.gov/large-docs/65/NCT07026565/ICF_001.pdf